CLINICAL TRIAL: NCT00430456
Title: Treadmill Exercise Prescriptions to Improve Fitness Versus Ambulatory Function After Stroke
Acronym: STEPs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H26843
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
Keywords: Aerobic exercise; Balance, postural; Cardiovascular deconditioning; Gait; MRI, functional; Physical therapy techniques; Self Efficacy; Treadmill test
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other): Higher Intensity, Shorter Duration Treadmill Training
  Interventions: Procedure: Exercise
- Arm 2 (Active Comparator): Lower Intensity, Longer Duration Treadmill Training
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — Treadmill Training

SUMMARY:
Individuals disabled by stroke are at risk of losing cardiovascular fitness and muscle due to disease. This worsens disability and can increase the risk of having another stroke or a heart attack. We would like to find out if and how different types of regular exercise (intense walking, long walking) can increase fitness, balance and improve walking function and activities of daily living in individuals who have suffered a stroke.

DETAILED DESCRIPTION:
This randomized study compares effects of duration vs. velocity-based TM training regimens on fitness and ambulatory function in chronic stroke patients. Phase 1 - patients are screened (Mini Mental Status, CESD for depression, alcohol intake survey) and undergo routine medical and CV evaluations and blood labs in VA RRDC Assessment Clinic to establish medical eligibility. Standard neurological evaluations (NIH Stroke Scale, Modified Asworth Spasticity Scale, range of motion and manual motor testing) and review of imaging records assess neurological eligibility, deficit profiles and stroke subtypes. Physician supervised treadmill tolerance test and peak effort constant velocity exercise stress test with vital signs monitoring determine treadmill safety, functional eligibility to participate (must walk 3 minutes at 0.2 MPH with handrail support), and cardiopulmonary safety in response to strenuous exertion. Eligible candidates undergo baseline testing (phase 2) including measures of fitness (VO2 peak, gait economy), ambulatory function and BOLD fMRI of knee movement. Phase 3 - 6 months TM training with either velocity or duration based progression, followed by Phase 4 -repeat of fitness and ambulatory function tests after 3 months, and Phase 5 - repeat of all baseline tests after 6 months training

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke greater than or equal to 6 months prior in men or women ages 40- 85 yrs. Hemorrhagic stroke greater than or equal to one year prior in men or women ages 40-85 years.
2. Residual hemiparetic gait deficits.
3. Already completed all conventional inpatient and outpatient physical therapy.
4. Adequate language and neurocognitive function to participate in exercise testing and training (specific screening instruments used.)

Exclusion Criteria:

1. Already performing aerobic exercise 3 X / week.
2. Increased alcohol consumption.
3. Cardiac history of:

   * unstable angina,
   * recent (less than 3 months) myocardial infarction, congestive heart failure (NYHA category II-IV);
   * hemodynamically significant valvular dysfunction.
4. Medical History:

   * recent hospitalization (less than 3 months) for severe medical disease,
   * PAOD with claudication,
   * orthopedic or chronic pain condition restricting exercise, pulmonary or renal failure,
   * active cancer,
   * untreated poorly controlled hypertension measured on at least 2 occasions ( greater than160/100) or diabetes mellitus (fasting glucose greater than 180 mg/dl, HgA1C greater than 10%) unable to be controlled medically within 3 months; g) Anemia defined by hematocrit less than 30 . (5) Neurological history of
   * dementia with Mini-Mental Status Score less than 23 (less than 17 if education level at or below 8th grade), and diagnostic confirmation by neurologist or psychiatrist,
   * severe receptive or global aphasia which confounds testing and training, operationally defined as unable to follow 2 point commands,
   * hemiparetic gait from a prior stroke preceding the index stroke defining eligibility,
   * non-stroke neuromuscular disorder restricting exercise (e.g. Parkinson's Syndrome),
   * untreated major depression. (6) BMI > 40.

Special fMRI Exclusion Criteria:

1. Metallic implants above the waist, except sternal wire implants.
2. Any type of implanted stimulator(cardiac, spinal, bladder, auditory
3. Claustrophobia
4. Pregnancy- A negative urine pregnancy test will be required prior to undergoing fMRI for women of child- bearing potential.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-08; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Peak Aerobic Fitness | 3 and 6 months

SECONDARY OUTCOMES:
Economy of Gait | 3 and 6 months
6 minute walk | 3 and 6 months
Fastest Comfortable 10-meter walk | 3 and 6 months
Self-Selected 10-meter walk | 3 and 6 months
48-hour Step Activity Monitoring | 3 and 6 months
Scales of Mobility, Function, Fatigue and Self-Efficacy | 6 months
Neuroplasticity (BOLD fMRI) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fred Ivey, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States